CLINICAL TRIAL: NCT00067041
Title: A Randomized Placebo-Controlled, 12-Week Multicenter Study of the Safety and Efficacy of Remodulin in Patients With Critical Limb Ischemia Following an Autogenous Vein Infrainguinal Bypass Graft
Brief Title: Effects of Remodulin in Patients With Critical Limb Ischemia Following a Vein Bypass Graft
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REM03:203
Record Dates: First submitted 2003-08-08; First posted 2003-08-13 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral Vascular Disease
Keywords: Critical Limb Ischemia; Autogenous Bypass Graft; CLI
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — treprostinil; Injections

INTERVENTIONS:
Drug: Remodulin (treprostinil sodium) Injection

SUMMARY:
Approximately 30 patients will be enrolled in this 12-week study designed to assess the effect of continuous subcutaneous Remodulin therapy on the outcome of infrainguinal bypass grafts in patients with critical limb ischemia (CLI). Portions of the study will be conducted in the hospital and on an out-patient basis. The study will be conducted at multiple centers.

ELIGIBILITY:
* Patients with critical limb ischemia and an appropriate reference lower-limb ischemic wound due to documented peripheral arterial disease who have had an autogenous vein infrainguinal bypass graft performed immediately prior to study initiation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-03; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Massachusetts Memorial Health Center, Worcester, Massachusetts
  - Vascular Institute Albany Medical College, Albany, New York
  - Oregon Health Sciences University, Portland, Oregon